CLINICAL TRIAL: NCT02855528
Title: Ultra Low-dose Coronary Artery Calcium Scoring Using Tin Filtration With Dual-source CT
Brief Title: Tin Filter Calcium Scoring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00051523
Record Dates: First submitted 2016-07-28; First posted 2016-08-04 (Estimated); Last update posted 2018-08-02 (Actual); Status verified 2018-03

CONDITIONS: Radiation Dose Reduction
Keywords: Tin Filter; Coronary Artery Calcium Scoring; Radiation dose reduction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Reduction of radiation dose and diagnostic accuracy (Experimental): Reduction of radiation dose during coronary artery calcium scoring with the use of a tin filter system.
  Interventions: Device: Tin Filter

INTERVENTIONS:
Device: Tin Filter

SUMMARY:
The aim of this study is to prospectively investigate the diagnostic performance and potential radiation dose reduction in coronary artery calcium scoring using the new tin filter system of the 3rd generation DSCT scanner.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be between 19-90 years of age.
* Subject must have been referred for a clinically indicated coronary artery calcium scan and/or coronary CT angiography or TRO scan with coronary artery calcium scoring.
* Subject must provide written informed consent prior to any study-related procedures being performed.
* Subject must be willing to comply with all clinical study procedures.

Exclusion Criteria:

* Subject is a pregnant or nursing female. Exclude the possibility of pregnancy:
* By testing (urine BHCG) within 24 hours before scan, or
* By surgical sterilization, or
* Post menopausal, with minimum one (1) year history without menses.
* Subject has an acute psychiatric disorder or is cognitively impaired.
* Subject is using or is dependent on substances of abuse.
* Subject is unwilling to comply with the requirements of the protocol.
* Subject is in acute unstable condition.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2015-12; Primary Completion 2017-11-14 (Actual); Study Completion 2017-11-14 (Actual)

PRIMARY OUTCOMES:
Reduction in radiation dose using the new tin-filter system | 2 years
Diagnostic accuracy of novel ultralow-dose non-enhanced coronary artery calcium scoring performed with the new tin filter system. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Joseph U. Schoepf, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States